CLINICAL TRIAL: NCT00356005
Title: Azithromycin Combination Therapy for the Treatment of Uncomplicated Falciparum Malaria in Bangladesh: An Open Label Randomized Controlled Trial
Brief Title: Azithromycin Combination Therapy for the Treatment of Uncomplicated Falciparum Malaria in Bangladesh
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Armed Forces Research Institute of Medical Sciences, Thailand (Other Government)
Responsible Party: Principal Investigator, Harald Noedl, Assoc. Prof., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICDDRB #2006-024; MUW #218/2006
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Uncomplicated Falciparum Malaria
Keywords: falciparum malaria; therapy; azithromycin; artesunate; Coartem; Bangladesh
MeSH Terms: conditions — Malaria, Falciparum | interventions — Azithromycin; Artesunate

ARMS (2):
- Azithromycin + Artesunate (Experimental): Azithromycin + Artesunate treatment
  Interventions: Drug: azithromycin plus artesunate
- Artesunate (Active Comparator): Artesunate treatment controls
  Interventions: Drug: Artesunate

INTERVENTIONS:
Drug: azithromycin plus artesunate
  Arms: Azithromycin + Artesunate
Drug: Artesunate
  Arms: Artesunate

SUMMARY:
The purpose of this study is to investigate the efficacy of azithromycin combination therapy with artesunate for the treatment of uncomplicated falciparum malaria in Bangladesh.

DETAILED DESCRIPTION:
In view of spreading antimalarial drug resistance there is an urgent need for new combination treatments for a disease that kills more than one million people every year. Azithromycin is a macrolide antibiotic that is particularly attractive due to its safety in children and experience with use in pregnancy. Recent trials suggest that azithromycin has a strong potential as an antimalarial. The purpose of this study is to investigate the efficacy of azithromycin combination therapy for the treatment of uncomplicated falciparum malaria in Bangladesh.

ELIGIBILITY:
Inclusion Criteria:

1. Acute symptomatic falciparum malaria infection with a parasite density of 100 to 100,000 asexual parasites/uL as determined on the screening smear with fever (defined as ≥37.5ºC), or reported history of fever within the last 48 hours.
2. Age: 8-65 years old
3. Males or females. All females over the age of 12 are required to have a negative human chorionic gonadotropin (hCG) pregnancy test (urine). All females of childbearing potential (not surgically sterile, or less than two years menopausal) are required to use an acceptable method of contraception, such as implant, injectable, oral contraceptive(s) with additional barrier contraception, intrauterine device, sexual abstinence, or vasectomized partner, throughout the study
4. Written informed consent obtained
5. Willing to stay under close medical supervision for the study duration
6. Otherwise healthy outpatients

Exclusion Criteria:

1. Pregnant women, nursing mothers, or women of childbearing potential who do not use an acceptable method of contraception (as described in Inclusion Criteria, #3)
2. Mixed malaria infection on admission by malaria smear
3. A previous history of intolerance or hypersensitivity to the study drugs artesunate, azithromycin, or lumefantrine or to drugs with similar chemical structures
4. Malaria drug therapy administered in the past 30 days by history
5. Previous participation in this trial, or participation in any other studies involving investigational or marketed products, concomitantly or within 30 days prior to entry in the study
6. History of significant cardiovascular, liver or renal functional abnormality or any other clinically significant illness, which in the opinion of the investigator would place them at increased risk.
7. Symptoms of severe vomiting (no food or inability to take food during the previous 8 hours).
8. Signs or symptoms of severe malaria (as defined by WHO 2003)
9. Unable and/or unlikely to comprehend and/or follow the protocol

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2006-08; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Primary clinical outcome is cure (ACPR as defined by WHO criteria) on Day 42. | 42 days

SECONDARY OUTCOMES:
Secondary outcome measures are time until parasite, fever, and gametocyte clearance (PCT, FCT, and GCT). | 42

CONTACTS AND LOCATIONS:
Overall Officials: Rashidul Haque, MBBS,PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh; Harald Noedl, MD, MCTM,PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Sadar Hospital, Bāndarban, Bangladesh

REFERENCES:
- [Derived] Thriemer K, Starzengruber P, Khan WA, Haque R, Marma AS, Ley B, Vossen MG, Swoboda P, Akter J, Noedl H. Azithromycin combination therapy for the treatment of uncomplicated falciparum malaria in Bangladesh: an open-label randomized, controlled clinical trial. J Infect Dis. 2010 Aug 15;202(3):392-8. doi: 10.1086/653710. PMID 20557237